CLINICAL TRIAL: NCT04088058
Title: Adipose-Derived Stem Cells (ADSCs) Injections for Liver Cirrhosis
Brief Title: A Phase II Open-label Single-arm Study to Evaluate the Efficacy and Safety of ADSCs in Subjects With Liver Cirrhosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gwo Xi Stem Cell Applied Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GXHPC1
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GXHPC1 (Experimental): One milliliter of cell suspension will be injected intrahepatically under sonographic guidance using a gauge-18 needle.
  Interventions: Drug: GXHPC1

INTERVENTIONS:
Drug: GXHPC1 — autologous ADSCs
  Other Names: hADSCs

SUMMARY:
The aim of the investigators study was to investigate the safety and efficacy of autologous ADSCs for the clinical treatment of liver cirrhosis.

DETAILED DESCRIPTION:
One milliliter of cell suspension will be injected intrahepatically under sonographic guidance using a gauge-18 needle.

ELIGIBILITY:
Inclusion Criteria:

Of either gender aged 20 to 70 years old (inclusive) 2. Diagnosed liver cirrhosis by CT imaging, irrespective of etiology 3. With MELD score 10 to 20 (inclusive) and Child-Pugh score 7 to 9 Note: MELD = Model For End-Stage Liver Disease 4. Subject with alcoholic cirrhosis should have been alcohol-abstinent for at least 6 months judged by psychiatrist with records for each month and willing to continue up to the completion of study.

5. Subject with cirrhosis caused by hepatitis B virus (HBV) should be with HBV DNA < 2,000 IU/mL before enrollment.

Note: HBV = hepatitis B virus, DNA = deoxyribonucleic acid. IU = International unit 6. Subject with cirrhosis caused by hepatitis C virus (HCV) should have successfully completed treatment for HCV with HCV viral load in the blood undetectable for at least 24 weeks since treatment cessation.

7. Provision of signed and dated informed consent form

Exclusion Criteria:

With inadequate coagulation function, as defined by: INR ≥ 1.5, aPTT ≥ 54.0 seconds, platelet count ≤ 50,000/mm3.

Note: INR = international normalized ratio, aPTT = activated partial thromboplastin time 2. With evidence of active autoimmune disease 3. With a medical record of malignancy within 5 years prior to screening, excluding curatively treated basal cell skin cancer, squamous cell skin cancer and carcinoma in situ of any site except urinary bladder.

4. With BMI ≤ 15 kg/m2 Note: BMI = body mass index 5. With inadequate hepatic function, as defined by: total bilirubin level > 5.0 mg/dL; AST > 3 × ULN, ALT > 3 × ULN, γ-GT > 4 × ULN, or ALP > 3 × ULN Note: γ-GT = Gamma-glutamyltransferase 6. With inadequate renal function, as defined by serum creatinine > 2.0 mg/dL The subject refuses to adopt highly effective contraceptives from signing informed consent to Final visit if female subject or female spouse/partner of male subject is of childbearing potential

Note: At least two forms of birth control must be adopted and one of which must be a barrier method. Acceptable forms of birth control include:

1. Established use of oral, injected or implanted hormonal methods of contraception
2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
3. Barrier methods of contraception: condom OR occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository 8. Female subject with childbearing potential who is pregnant (confirmed by urine or serum pregnancy test) or lactating 9. Having participated other investigational study within 4 weeks of entering this study 10. Has a known allergy to study intervention or its excipients. If there is suspicion that the subject may have an allergy, the subject should be excluded.

   11. With ongoing infection requiring systemic treatment such as HIV, syphilis or acute infectious disease except HBV or HCV Note: HIV = human immunodeficiency virus 12. With drug dependency for the past 1 year of Screening visit 13. With any rare diseases 14. With uncontrolled hypertension (≥180/≥110 mmHg on more than 2 antihypertensive medications) or uncontrolled diabetic mellitus (HbA1c > 9.0%) 15. With liver abscess or moderate to severe (or refractory) ascites 16. With uncontrolled psychiatric disorder or altered mental status precluding informed consent or necessary testing 17. Having received major surgery within past 12 weeks of Screening visit

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-16 (Actual); Primary Completion 2025-04-19 (Estimated); Study Completion 2025-04-19 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 48 in The METAVIR score | 48 weeks
  The METAVIR score is a tool used to evaluate the severity of fibrosis seen on a liver biopsy sample. The METAVIR score grades the degree of fibrosis on a 5-point scale from 0 to 4 as follows:
  F0: No fibrosis F1: Portal fibrosis without septa F2: Portal fibrosis with few septa F3: Numerous septa without cirrhosis F4: Cirrhosis

SECONDARY OUTCOMES:
Change from Baseline to Week 24 in The METAVIR score | 24 weeks
  The METAVIR score is a tool used to evaluate the severity of fibrosis seen on a liver biopsy sample. The METAVIR score grades the degree of fibrosis on a 5-point scale from 0 to 4 as follows:
  F0: No fibrosis F1: Portal fibrosis without septa F2: Portal fibrosis with few septa F3: Numerous septa without cirrhosis F4: Cirrhosis
Change from baseline to Weeks 24, and 48 in Fibroscan® score for liver elasticity | 24 weeks, 48 weeks
  Fibroscan® is a non-invasive modality to measure elasticity of liver tissue. A fibroscan® score is a numerical result between 2-75. A 'normal' Fibroscan range tends to be between 2-7 with an average result being roughly around 5. Scarring of the liver is measured by four stages.
  F0 = no scarring F1 = mild fibrosis F2 = moderate fibrosis F3 = severe fibrosis F4 = cirrhosis or advanced fibrosis
Change from baseline to Weeks 12, 24, 36, and 48 in the MELD score | 12 weeks, 24 weeks, 36 weeks, 48 weeks
  The Model for End-Stage Liver Disease, or MELD, is a scoring system for assessing the severity of the chronic liver disease. MELD score is calculated according to the subject's values for serum total bilirubin, serum creatinine, and INR.
Change from baseline to Weeks 12, 24, 36, and 48 in the Child-Pugh score | 12 weeks, 24 weeks, 36 weeks, 48 weeks
  The Child-Pugh score is used to assess the prognosis of chronic liver disease, mainly cirrhosis. The score employs five clinical measures of liver disease. Each measure is scored 1-3, with 3 indicating most severe derangement.
Incidence of adverse event(AE) and SAE | 0-48 weeks
  An adverse event (AE) can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not relate with the medicinal (investigational) product.
Incidence of serious adverse event (SAE) | 0-48 weeks
  An adverse event (AE) or suspected adverse reaction is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes (based on ICH
  GCP):
  * results in death,
  * is life-threatening,
  * requires inpatient hospitalization or prolongation of existing hospitalization,
  * results in persistent or significant disability/incapacity, or
  * is a congenital anomaly/birth defect

CONTACTS AND LOCATIONS:
Overall Officials: Huang ka Wen, Director, Principal Investigator — National Taiwan University Hospital; Lee Mi Che, Director, Principal Investigator — Hualien Tzu Chi General Hospital
Locations (2):
- Taiwan (2):
  - HualienTzu Chi Hospital, Hualien City
  - National Taiwan University Hospital, Taipei County